CLINICAL TRIAL: NCT07258641
Title: Dual Wavelength Fluorescence Imaging Using Fluorescently Labelled Adalimumab and Risankizumab for Visualizing Drug Targeting in Inflammatory Bowel Diseases
Brief Title: Fluorescence Imaging of Adalimumab-680LT and Risankizumab-800CW in Inflammatory Bowel Disease
Acronym: VOYAGER
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: UMCG 21773; 2025-521420-30-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-04

CONDITIONS: Ulcerative Colitis (UC); Crohn Disease (CD)
Keywords: Fluorescence Molecular Endoscopy; Inflammatory Bowel Disease; Risankizumab-800CW; Adalimumab-680LT
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 25 mg adalimumab-680LT and 15/25 mg risankizumab-800CW (Experimental): Patients receive 25 mg adalimumab-680LT and 15/25 mg risankizumab-800CW and undergo a Fluorescence Molecular Imaging Procedure
  Interventions: Drug: 25mg adalimumab-680LT and 15/25 mg risankizumab-800CW
- 25 mg adalimumab-680LT (Experimental): Patients starting with adalimumab will receive 25 mg adalimumab-680LT and undergo a Fluorescence Molecular Imaging procedure
  Interventions: Drug: Adalimumab-680LT 25mg
- 15/25 mg risankizumab-800CW (Experimental): Patients starting with risankizumab receive 15/25 mg risankizumab-800CW and undergo a Fluorescence Molecular Imaging procedure
  Interventions: Drug: Risankizumab-800CW 15 mg/25 mg
- No second procedure (No Intervention): Patients starting with drugs other than adalimumab or risankizumab will not undergo a second procedure

INTERVENTIONS:
Drug: 25mg adalimumab-680LT and 15/25 mg risankizumab-800CW — Adalimumab-680LT and risankizumab-800CW will be administered intravenously. 2-3 days later, a Fluorescence Molecular Imaging procedure will be performed to enable the visualisation and detection of dual-wavelength fluorescence signals.
  Arms: 25 mg adalimumab-680LT and 15/25 mg risankizumab-800CW
Drug: Adalimumab-680LT 25mg — Adalimumab-680LT will be administered intravenously. 2-3 days later, a Fluorescence Molecular Imaging procedure will be performed to enable the visualisation and detection of fluorescence signals.
  Arms: 25 mg adalimumab-680LT
Drug: Risankizumab-800CW 15 mg/25 mg — Risankizumab-800CW will be administered intravenously. 2-3 days later, a Fluorescence Molecular Imaging procedure will be performed to enable the visualisation and detection of fluorescence signals.
  Arms: 15/25 mg risankizumab-800CW

SUMMARY:
Inflammatory bowel diseases (IBD) are chronic relapsing inflammatory disorders of the gastrointestinal tract affecting 2.5 million patients in Europe alone. The majority of newly diagnosed patients are in adolescence or early adulthood and in the midst of their family life, career, and social development.

IBD comes with significant morbidity and complex treatment strategies and is associated with a high social burden and medical costs. Besides other factors, the pathogenesis of IBD is attributed to proinflammatory cytokine tumor necrosis factor α (TNFα) and Interleukin 23 (IL-23). Adalimumab, a human monoclonal anti-TNF antibody, and risankizumab, a humanized monoclonal anti-IL-23 antibody, are used to treat patients with moderate to severely active IBD. However, IBD patients often only partially respond to such biological immunomodulating therapies, resulting in high primary nonresponse (30-60%) and loss of response over time (48-58%). The investigators are currently missing reliable tools for response prediction because the limitations of current technologies do not allow the visualization of the molecular phenotype or heterogeneity within patients. Therefore, patients are potentially exposed to a non-effective treatment and its potential side effects while clinical deterioration is ongoing. In addition, it remains completely unknown for most biologicals used for IBD therapy whether they reach their actual targets in the tissue and if a sufficient local concentration is present to achieve treatment response. To develop a predictive tool for assessment of therapeutic (non-)response to patients and gain insights into local drug concentrations in individual patients before initiating anti-TNF or anti-IL23 therapy, the University Medical Center Groningen (UMCG), fluorescently labeled adalimumab (adalimumab-680LT) and risankizumab (risankizumab-800CW) to visualize and quantify the labeled drugs in diseased tissue with dedicated optical fluorescence imaging systems. In previous studies, the investigators have proven that those tracers bind to TNFα/IL23 in the mucosa after intravenous injection and that the investigators can investigate the drug distribution in vivo due to the colocalization of the fluorescently labeled compound. The aim of this follow-up study is to assess the feasibility of simultaneous dual wavelength imaging of adalimumab-680LT and risankizumab-800CW at baseline and evaluate target saturation after at least 14 weeks of adalimumab or risankizumab therapy. The investigators will also use in vivo and ex vivo fluorescence molecular imaging (FMI) to visualize tracer target cells and the patient's molecular phenotype for potential treatment response prediction in IBD patients in the future.

The investigators will determine the feasibility of dual wavelengths molecular fluorescence imaging using the GMPproduced near-infrared fluorescent tracers adalimumab-680LT and risankizumab-800CW for visualizing medicine distribution in and ex vivo IBD patients with dedicated fluorescence imaging systems.

Furthermore, the investigators will evaluate TNF and IL23 target saturation after 14 weeks of adalimumab or risankizumab therapy and characterize the tissue microenvironment where the drug is abundant and identify potential drug target cells.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion meet all of the following criteria:

* Established IBD diagnosis (UC or CD).
* Active disease: clinically active disease of the bowel is defined as at least mild activity using dedicated scoring indices or biochemically active disease as defined by a fecal calprotectin > 60 µg/g
* Patients must be eligible for adalimumab or risankizumab therapy.
* Age of 18 years
* Written informed consent
* Clinical indication for an endoscopic procedure

For female subjects who are of childbearing potential, are premenopausal with intact reproductive organs, or are less than 2 years postmenopausal:

• A negative pregnancy test (urine or blood test) must be available.

Exclusion Criteria:

A female study patient who is pregnant or provides breastfeeding

* A female study patient of premenopausal age who does not use any reliable form of contraception at the time of adalimumab-680LT and/or risankizumab 800CW administration
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent
* Prior anti-IL23-specific therapy (IL23/IL12 combination therapy is not an exclusion criteria)
* Prior anti-TNFα therapy in the last 6 weeks before inclusion
* Previous treatment with adalimumab and detectable anti-adalimumab antibody levels

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
To investigate the feasibility of using dual wavelengths fluorescence molecular endoscopy (FME) | 12 months
  Visual evaluation and distinction of both tracers during FME (visible signal yes/no), as well as TBR and CNR calculations, will be performed to assess in vivo signal detectability.
To investigate the feasibility of using ex vivo fluorescence molecular imaging (FMI) to detect adalimumab-680LT and risankizumab-800CW signals | 12 months
  Ex vivo analysis will include mean fluorescence intensities (MFIs) of biopsies, MDSFR/SFF measurements, and fluorescence and light sheet microscopy to quantify and localize tracer signals.
Blood pressure | Five minutes before, and five and sixty minutes after tracer administration
  Systolic and diastolic in millimeters of mercure (mmHg)
Heart rate | Five minutes before, and five and sixty minutes after tracer administration
  Beats per minute
Temperature | Five minutes before, and five and sixty minutes after tracer administration
  Degrees Celsius

SECONDARY OUTCOMES:
To investigate a potential correlation of in vivo and ex vivo fluorescence signal intensities and target saturation to clinical response/remission after 14 weeks of adalimumab/risankizumab therapy regimen in patients with IBD. | 12 months
  This will involve semi-quantitative and spectroscopic analysis of fluorescence signals during endoscopy and in biopsies, comparison with inflammation scores, and molecular validation of tracer binding and immune cell localization to assess predictive and response-related biomarkers.
To quantify the fluorescence signals of the tracers in vivo by using single-fiber reflectance/single-fiber fluorescence (MDSFR/SFF) spectroscopy and correlate these measurements to inflammation severity. | 12 months
  This will be achieved through real-time spectroscopic quantification of fluorescence signals during endoscopy in each investigated bowel segment, followed by comparison with endoscopic and histologic inflammation scores to assess the relationship between tracer signal intensity and tissue inflammation.
To evaluate the adalimumab-680LT and risankizumab-800CW distribution inside mucosal biopsies | 12 months
  This will be achieved through 3D ex vivo fluorescence signal analysis of intact biopsies collected from high and low fluorescence areas during endoscopy, enabling assessment of tracer distribution across inflamed and non-inflamed tissue. Additional validation will include SDS-PAGE to confirm tracer integrity, fluorescence microscopy, and immunofluorescence staining to visualize and quantify tracer-positive cells and their immune cell types.
To identify the composition of immune cells in the mucosal microenvironment of IBD patients and gain new insights into the target cells and distribution of adalimumab and risankizumab | 12 months
  This will be addressed through fluorescence microscopy and immunofluorescence staining of FFPE biopsy slides to visualize adalimumab-680LT and risankizumab-800CW signals and identify immune cell types (e.g., CD68, CD3, CD8, CD20). The number and distribution of tracer-positive cells and immune subsets will be quantified to explore associations with therapy response and mucosal immune profiles.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No